CLINICAL TRIAL: NCT06385873
Title: Disitamab Vedotin Combined With Adebrelimab, Apatinib and S-1 as Neoadjuvant Therapy in Locally Advanced Gastric Cancer With HER2 Overexpression: a Prospective, Phase II Study
Brief Title: RC48 Combined With Adebrelimab, Apatinib and S-1 as Neoadjuvant Therapy in Locally Advanced Gastric Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-SR-233
Record Dates: First submitted 2024-04-24; First posted 2024-04-26 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer/Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — disitamab vedotin; apatinib; S 1 (combination); gimeracil; potassium oxonate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): RC48, Adebrelimab, Apatinib and S-1 regimen for 3-4 cycles (every 3 weeks) before surgery.
  Interventions: Drug: RC48; Drug: Adebrelimab; Drug: Apatinib; Drug: S-1

INTERVENTIONS:
Drug: RC48 — RC48: 2.5 mg/kg, intravenous infusion, on day 1, every 3 weeks (Q3W);
  Other Names: Disitamab Vedotin
Drug: Adebrelimab — Adebrelimab：1200 mg, intravenous infusion, on day 1, every 3 weeks (Q3W);
Drug: Apatinib — Apatinib: 250mg, oral administration, once daily (qd), every 3 weeks (Q3W);
Drug: S-1 — S-1：For patients with a body surface area (BSA) ≤1.5m², use 50mg each time; for patients with BSA >1.5m², use 60mg each time, oral administration, twice daily (bid), on days 1-14, every 3 weeks (Q3W);
  Other Names: S-1tegafur, gimeracil and oteracil potassium

SUMMARY:
This study is a prospective, open-label, phase II clinical trial that aims to enroll patients with locally advanced gastric adenocarcinoma who have not received any prior treatment and are candidates for surgery. The study drugs include RC48, Adebrelimab, Apatinib and S-1. The purpose is to evaluate the effectiveness and safety of the combined coordinated treatment of multi-mechanism drugs for perioperative treatment of locally advanced gastric cancer with HER2 overexpression.

DETAILED DESCRIPTION:
The study plans to enroll 32 subjects. After signing the informed consent form and meeting the inclusion and exclusion criteria, patients will receive standard-dose treatment of the RC48, Adebrelimab, Apatinib and S-1 regimen for 3-4 cycles (every 3 weeks) before surgery. Apatinib will only be used for 14 days in the last cycle. Imaging studies will be conducted 3-4 weeks after the last dose to assess the efficacy of neoadjuvant therapy and the possibility of radical D2 gastrectomy. The treatment plan after curative surgery for gastric cancer will be determined by the investigators and the patients based on the pathological findings. Patients who benefit clinically after surgery may receive adjuvant therapy with RC48, Adebrelimab, Apatinib and S-1 for 4 cycles (the first treatment is expected to start around 4 weeks after surgery) or follow the standard postoperative adjuvant regimen recommended by the guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 1. Participants voluntarily join this study, are able to complete the signing of the informed consent form, and have good compliance;
* 2. Age between 18 to 75 years old (at the time of signing the informed consent form), with no gender restrictions;
* 3. Gastrointestinal cancer or gastroesophageal junction adenocarcinoma confirmed by histology and/or cytology, diagnosed as locally advanced according to the 8th edition of the AJCC standards, with a cTNM diagnosis of T3-4aN+M0 and T4aNanyM0 based on ultrasound endoscopy or enhanced CT/MRI scan (and diagnostic laparoscopy if necessary), and agree to receive curative surgical treatment, with the investigator assessing the potential for tumor resectability;
* 4. Have not previously received systemic treatment for the current disease, including anti-tumor chemotherapy/immunotherapy, etc.;
* 5. HER2 overexpression confirmed by IHC results from endoscopic biopsy tissue (defined as: IHC 2+, 3+);
* 6. ECOG score of 0-1;
* 7. Estimated life expectancy of ≥6 months;
* 8. Good major organ function:

Exclusion Criteria:

* 1. Concurrent malignant disease other than gastric cancer (excluding early-stage tumors that have been radically treated);
* 2. Tumor lesions with a tendency to bleed (such as active ulcerative tumor lesions with positive fecal occult blood test, history of hematemesis or melena within 2 months before signing the informed consent form, or assessed by the investigator as being at risk of significant gastrointestinal hemorrhage, etc.) or having received blood transfusion treatment within 4 weeks before the study medication; 3. Inability to take oral medication;
* 4. Currently participating in another interventional clinical study treatment, or having received other investigational drugs or used investigational medical devices within 4 weeks before the first administration of the study medication;
* 5. Has had systemic treatment required within 2 years before the first administration of the study medication;
* 6. Known allogeneic organ transplantation (except for corneal transplantation);
* 7. Known allergy to any medication used in this study;
* 8. Peripheral neuropathy of grade ≥2;
* 9. Known history of human immunodeficiency virus (HIV) infection (i.e., positive for HIV 1/2 antibodies);
* 10. Active hepatitis B or C infection;
* 11. Received live vaccines within 30 days before the first administration (Day 1 of Cycle 1);
* 12. Pregnant or breastfeeding women;
* 13. Presence of any severe or uncontrollable systemic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response Rate (pCR) | 4 months
  Defined as the proportion of subjects with no residual viable tumor cells on microscopy and negative lymph nodes out of the total number of subjects;

SECONDARY OUTCOMES:
Major Pathological Response rate (MPR) | 4 months
  Defined as the proportion of subjects with ≤10% viable tumor cells in the resected specimen out of the total number of subjects;
R0 Resection rate | 4 months
  Complete tumor resection during surgery with negative microscopic margins, meaning no residual tumor;
Disease-Free Survival (DFS） | 24 months
  Defined as the time from enrollment to the first radiological evidence of disease recurrence or death (whichever occurs first)
Overall Survival (OS) | 36 months
  Defined as the time from enrollment to the subject's death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Xiaofeng, Ph.D, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Hao Xu, Ph.D, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University

IPD SHARING:
Plan to Share IPD: No